CLINICAL TRIAL: NCT05456529
Title: A Phase 3, Open-Label, One-Year Safety Study of Ruxolitinib Cream in Adolescents (Ages ≥ 12 Years to < 18 Years) With Atopic Dermatitis
Brief Title: Study of Ruxolitinib Cream in Adolescents With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-315
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis (AD)
Keywords: atopic dermatitis (AD); adolescents; pruritus; eczema; topical therapy; JAK inhibitor
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Ruxolitinib cream 1.5% twice daily (BID) during the continuous and LTS treatment period.
  Interventions: Drug: Ruxolitinib Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream 1.5% twice daily (BID) during the continuous and LTS treatment period.
  Other Names: INCB18424 cream

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of ruxolitinib cream in adolescents with Atopic Dermatitis (AD).

DETAILED DESCRIPTION:
The study comprises of a 8 week continuous treatment period followed by 44 week Long Term Safety (LTS) period and 30 days safety follow up period. During Continuous treatment period all lesions identified at baseline will be treated and during LTS period only active lesions will be treated.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Atopic Dermatitis (AD) as defined by the Hanifin and Rajka (1980) criteria.
* Duration of AD of at least 2 years.
* Total IGA score of 2 to 3 at the screening and baseline visits.
* Percent BSA (excluding the scalp) with AD involvement of 3% to 20% at the screening and baseline visits.
* Atopic dermatitis not adequately controlled with other topical prescription therapies or when those therapies are not advisable.
* Agree to discontinue all agents used to treat AD from screening through the final follow up visit.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* An unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to baseline.
* Concurrent conditions and history of other diseases
* Any current and/or history of serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including application of study cream and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data. For example:
* Clinically significant or uncontrolled cardiovascular disease, including unstable angina, acute myocardial infarction or stroke within 6 months from Day 1 of study cream application, New York Heart Association Class III or IV congestive heart failure, and arrhythmia requiring therapy or uncontrolled hypertension (blood pressure > 150/90 mm Hg) unless approved by the medical monitor/sponsor.
* Current and/or history of malignancy in the 5 years preceding the baseline visit, except for adequately treated, nonmetastatic nonmelanoma skin cancer.
* Current and/or history of arterial or venous thrombosis, including DVT and PE.
* Current and/or history of active tuberculosis or current and/or history of latent tuberculosis unless adequately treated.
* Any of the following clinical laboratory test results at screening:

  1. Hemoglobin < 100 g/L (< 10 g/dL)
  2. Liver function tests:
* AST or ALT ≥ 2.5 × ULN
* Total bilirubin > 1.5 × ULN with the exception of Gilbert disease. c. Estimated glomerular filtration rate < 30 mL/min/1.73 m2 (using the CKD Epidemiology Collaboration equation).

  d. Positive serology test results for HIV antibody. e. Any other clinically significant laboratory result that, in the opinion of the investigator, poses a significant risk to the participant.
* Use of any of the following treatments within the indicated washout period before baseline:

  1. 5 half-lives or 12 weeks, whichever is longer - biologic agents (eg, dupilumab).
  2. 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogues, cyclosporine, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (eg, mycophenolate or tacrolimus).
  3. 2 weeks - immunizations with live-attenuated vaccines; sedating antihistamines, unless on long-term stable regimen (nonsedating antihistamines are permitted).

     Note: Live-attenuated vaccines are not recommended during the CT period. Note: COVID-19 vaccination is allowed.
  4. 1 week - use of other topical treatments for AD (other than bland emollients, eg, Aveeno® creams, ointments, sprays, soap substitutes), such as topical antipruritics (eg, doxepin cream), corticosteroids, calcineurin inhibitors, PDE4 inhibitors, coal tar (shampoo), antibiotics, or antibacterial cleansing body wash/soap.

Note: Diluted sodium hypochlorite "bleach" baths are allowed as long as they do not exceed 2 baths per week and their frequency remains the same throughout the study.

* Previously received systemic or topical JAK inhibitors (eg, ruxolitinib, tofacitinib, baricitinib, filgotinib, lestaurtinib, pacritinib).
* Ultraviolet light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, sunlight or tanning booth) within 2 weeks prior to the baseline visit and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the participant's AD.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before baseline with another investigational medication or current enrollment in another investigational drug protocol.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before baseline with a strong CYP3A4 inhibitor.
* Inability to draw blood for PK analysis from any nonlesional areas.
* Known allergy or reaction to any component of the study cream formulation.
* In the opinion of the investigator unable or unlikely to comply with the administration schedule and study evaluations.

Further exclusion criteria may apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Angel, MD, Study Director — Incyte Corporation
Locations (38):
- United States (26):
  - Arkansas Research Trials, North Little Rock, Arkansas
  - First Oc Dermatology, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Peninsula Research Associates Pra, Rolling Hills Estates, California
  - Advanced Rx Clinical Research Group, Inc, Westminster, California
  - Encore Medical Research, Llc Hollywood, Hollywood, Florida
  - Solutions Through Advanced Research, Inc, Jacksonville, Florida
  - Acevedo Clinical Research, Miami, Florida
  - Skin Research of South Florida, Llc, Miami, Florida
  - Well Pharma Medical Research Corp., Miami, Florida
  - Forward Clinical Trials, Tampa, Florida
  - Iact Health, Columbus, Georgia
  - Sneeze Wheeze and Itch Associates Llc, Normal, Illinois
  - Northshore University Health System, Skokie, Illinois
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - Skin Specialists Pc the Advanced Skin Research Center, Omaha, Nebraska
  - Empire Dermatology, East Syracuse, New York
  - Sadick Dermatology Sadick Research Group, New York, New York
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Aventiv Research Inc-Dublin, Dublin, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Arlington Research Center, Arlington, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Jordan Valley Medical Center, West Jordan, Utah
- Canada (6):
  - Dermatology Research Institute, Calgary, Alberta
  - Dr. Chih-Ho Hong Medical Inc., Surrey, British Columbia
  - Lmc Manna Research (London), London, Ontario
  - Manna Research Toronto, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Xlr8 Medical Research, Windsor, Ontario
- Poland (6):
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Centrum Medyczne Angelius Provita, Katowice
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Dermedic Dr. Zdybski, Ostrowiec Świętokrzyski
  - Centrum Medyczne Evimed, Warsaw
  - Klinika Ambroziak, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 25 study centers in the United States and Canada.
Groups:
- Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) to all areas identified for treatment at Baseline regardless of whether or not the lesion(s) improved for 8 weeks (Continuous Treatment Period). Participants who completed the Week 8 assessments with no safety concerns and with a percentage of body surface area (%BSA) affected by atopic dermatitis of no greater than 20% continued into the Long-term Safety (LTS) Period. During the 44 weeks of the LTS Period, the treatment regimen continued to be ruxolitinib 1.5% cream BID; however, participants only treated active atopic dermatitis lesions.
Period: 8-week Continuous Treatment (CT) Period
Arm/Group | Ruxolitinib 1.5% Cream BID
Started | 103
Completed | 92
Not Completed | 11
Not completed — Lost to Follow-up | 5
Not completed — Lack of Efficacy | 2
Not completed — Protocol-specified Withdrawal Criterion Met | 1
Not completed — Withdrawal by Subject | 3
Period: 44-week Long-term Safety Period
Arm/Group | Ruxolitinib 1.5% Cream BID
Started | 92
Completed | 61
Not Completed | 31
Not completed — Lost to Follow-up | 12
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 2
Not completed — Protocol-specified Withdrawal Criterion Met | 1
Not completed — Withdrawal by Subject | 12
Not completed — Withdrawal by Sponsor | 2
Not completed — Unable to Attend the Follow-up Visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 80
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 46
  Black/African-American | 31
  Asian | 18
  Native Hawaiian/Pacific Islander | 2
  Unknown | 1
  Asian/White | 1
  Middle Eastern (Arab) | 1
  East Indian | 1
  White/Black | 1
  Asian, Dominican, Cuban | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study cream. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first application of study cream and up to 30 days after the last application of study cream.
Time Frame: up to 462 days
Population: Full Analysis Set: all participants who applied ruxolitinib cream at least once
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants | 42

2. Primary Outcome: Number of Participants With ≥Grade 3 TEAEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was drug related. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first application of study cream and up to 30 days after the last application of study cream. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 462 days
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants | 3

3. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Basophil, Eosinophil, Leukocyte, Lymphocyte, Monocyte, Neutrophil, and Platelet Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils, and platelets were measured in 10^9 cells per liter.
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Basophils, low | 0
  Basophils, normal | 94
  Basophils, high | 1
  Basophils, low and high | 0
  Basophils, missing | 8
  Eosinophils, low | 0
  Eosinophils, normal | 83
  Eosinophils, high | 19
  Eosinophils, low and high | 0
  Eosinophils, missing | 1
  Leukocytes, low | 18
  Leukocytes, normal | 83
  Leukocytes, high | 1
  Leukocytes, low and high | 0
  Leukocytes, missing | 1
  Lymphocytes, low | 7
  Lymphocytes, normal | 95
  Lymphocytes, high | 0
  Lymphocytes, low and high | 0
  Lymphocytes, missing | 1
  Monocytes, low | 0
  Monocytes, normal | 92
  Monocytes, high | 10
  Monocytes, low and high | 0
  Monocytes, missing | 1
  Neutrophils, low | 13
  Neutrophils, normal | 87
  Neutrophils, high | 2
  Neutrophils, low and high | 0
  Neutrophils, missing | 1
  Platelets, low | 5
  Platelets, normal | 75
  Platelets, high | 21
  Platelets, low and high | 1
  Platelets, missing | 1

4. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Baso/Leuko, Eosino/Leuko, Lymphocyte/Leuko, Monocyte/Leuko, and Neutro/Leuko Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Basophils (baso)/leukocytes (leuk), eosinophils (eosino)/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes, and neutrophils (neutro)/leukocytes were measured as a percentage.
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Basophils/leukocytes, low | 0
  Basophils/leukocytes, normal | 84
  Basophils/leukocytes, high | 18
  Basophils/leukocytes, low and high | 0
  Basophils/leukocytes, missing | 1
  Eosinophils/leukocytes, low | 0
  Eosinophils/leukocytes, normal | 73
  Eosinophils/leukocytes, high | 29
  Eosinophils/leukocytes, low and high | 0
  Eosinophils/leukocytes, missing | 1
  Lymphocytes/leukocytes, low | 29
  Lymphocytes/leukocytes, normal | 47
  Lymphocytes/leukocytes, high | 22
  Lymphocytes/leukocytes, low and high | 4
  Lymphocytes/leukocytes, missing | 1
  Monocytes/leukocytes, low | 3
  Monocytes/leukocytes, normal | 94
  Monocytes/leukocytes, high | 5
  Monocytes/leukocytes, low and high | 0
  Monocytes/leukocytes, missing | 1
  Neutrophils/leukocytes, low | 6
  Neutrophils/leukocytes, normal | 66
  Neutrophils/leukocytes, high | 30
  Neutrophils/leukocytes, low and high | 0
  Neutrophils/leukocytes, missing | 1

5. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Erythrocyte Mean Corpuscular Volume and Mean Platelet Volume Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Erythrocyte mean corpuscular volume and mean platelet volume were measured in femtoliters.
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Erythrocyte mean corpuscular volume, low | 3
  Erythrocyte mean corpuscular volume, normal | 88
  Erythrocyte mean corpuscular volume, high | 11
  Erythrocyte mean corpuscular volume, low and high | 0
  Erythrocyte mean corpuscular volume, missing | 1
  Mean platelet volume, low | 5
  Mean platelet volume, normal | 97
  Mean platelet volume, high | 0
  Mean platelet volume, low and high | 0
  Mean platelet volume, missing | 1

6. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Erythrocyte Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Erythrocytes were measured in 10^12/Liter.
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Low | 14
  Normal | 66
  High | 22
  Low and high | 0
  Missing | 1

7. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Hematocrit Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Hematocrit was measured in liters of red blood cells per liter of blood (L/L).
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Low | 2
  Normal | 88
  High | 12
  Low and high | 0
  Missing | 1

8. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Hemoglobin Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Hemoglobin was measured in grams per liter.
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Low | 19
  Normal | 79
  High | 4
  Low and high | 0
  Missing | 1

9. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Basophil, Eosinophil, Leukocyte, Lymphocyte, Monocyte, Neutrophil, and Platelet Value of Low, Normal, High, Low and High, and Missing
Description: as for outcome 3
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: Long-term Safety (LTS) Evaluable Population: all participants who applied ruxolitinib cream at least once during the LTS Period
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Basophils, low | 0
  Basophils, normal | 85
  Basophils, high | 2
  Basophils, low and high | 0
  Basophils, missing | 5
  Eosinophils, low | 0
  Eosinophils, normal | 63
  Eosinophils, high | 25
  Eosinophils, low and high | 0
  Eosinophils, missing | 4
  Leukocytes, low | 20
  Leukocytes, normal | 62
  Leukocytes, high | 6
  Leukocytes, low and high | 0
  Leukocytes, missing | 4
  Lymphocytes, low | 5
  Lymphocytes, normal | 82
  Lymphocytes, high | 1
  Lymphocytes, low and high | 0
  Lymphocytes, missing | 4
  Monocytes, low | 0
  Monocytes, normal | 75
  Monocytes, high | 13
  Monocytes, low and high | 0
  Monocytes, missing | 4
  Neutrophils, low | 12
  Neutrophils, normal | 66
  Neutrophils, high | 10
  Neutrophils, low and high | 0
  Neutrophils, missing | 4
  Platelets, low | 3
  Platelets, normal | 60
  Platelets, high | 25
  Platelets, low and high | 0
  Platelets, missing | 4

10. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Baso/Leuko, Eosino/Leuko, Lymphocyte/Leuko, Monocyte/Leuko, and Neutro/Leuko Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Basophils (baso)/leukocytes (leuko), eosinophils (eosino)/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes, and neutrophils (neutro)/leukocytes were measured as a percentage.
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Basophils/leukocytes, low | 0
  Basophils/leukocytes, normal | 67
  Basophils/leukocytes, high | 21
  Basophils/leukocytes, low and high | 0
  Basophils/leukocytes, missing | 4
  Eosinophils/leukocytes, low | 0
  Eosinophils/leukocytes, normal | 49
  Eosinophils/leukocytes, high | 39
  Eosinophils/leukocytes, low and high | 0
  Eosinophils/leukocytes, missing | 4
  Lymphocytes/leukocytes, low | 39
  Lymphocytes/leukocytes, normal | 29
  Lymphocytes/leukocytes, high | 18
  Lymphocytes/leukocytes, low and high | 2
  Lymphocytes/leukocytes, missing | 4
  Monocytes/leukocytes, low | 13
  Monocytes/leukocytes, normal | 68
  Monocytes/leukocytes, high | 7
  Monocytes/leukocytes, low and high | 0
  Monocytes/leukocytes, missing | 4
  Neutrophils/leukocytes, low | 8
  Neutrophils/leukocytes, normal | 43
  Neutrophils/leukocytes, high | 37
  Neutrophils/leukocytes, low and high | 0
  Neutrophils/leukocytes, missing | 4

11. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Erythrocyte Mean Corpuscular Volume and Mean Platelet Volume Value of Low, Normal, High, Low and High, and Missing
Description: as for outcome 5
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Erythrocyte mean corpuscular volume, low | 4
  Erythrocyte mean corpuscular volume, normal | 56
  Erythrocyte mean corpuscular volume, high | 28
  Erythrocyte mean corpuscular volume, low and high | 0
  Erythrocyte mean corpuscular volume, missing | 4
  Mean platelet volume, low | 11
  Mean platelet volume, normal | 77
  Mean platelet volume, high | 0
  Mean platelet volume, low and high | 0
  Mean platelet volume, missing | 4

12. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Erythrocyte Value of Low, Normal, High, Low and High, and Missing
Description: as for outcome 6
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Low | 19
  Normal | 42
  High | 26
  Low and high | 1
  Missing | 4

13. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Hematocrit Value of Low, Normal, High, Low and High, and Missing
Description: as for outcome 7
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Low | 2
  Normal | 49
  High | 37
  Low and high | 0
  Missing | 4

14. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Hemoglobin Value of Low, Normal, High, Low and High, and Missing
Description: as for outcome 8
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Low | 26
  Normal | 55
  High | 7
  Low and high | 0
  Missing | 4

15. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline ALT, ALP, AST, CL, and LDH Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Alanine aminotransferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST), creatine kinase (CK), and lactate dehydrogenase (LDH) were measured in units per liter.
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  ALT, low | 0
  ALT, normal | 100
  ALT, high | 3
  ALT, low and high | 0
  ALT, missing | 0
  ALP, low | 14
  ALP, normal | 89
  ALP, high | 0
  ALP, low and high | 0
  ALP, missing | 0
  AST, low | 0
  AST, normal | 102
  AST, high | 1
  AST, low and high | 0
  AST, missing | 0
  CK, low | 3
  CK, normal | 77
  CK, high | 22
  CK, low and high | 1
  CK, missing | 0
  LDH, low | 7
  LDH, normal | 91
  LDH, high | 5
  LDH, low and high | 0
  LDH, missing | 0

16. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Albumin Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Albumin was measured in grams per liter.
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Low | 0
  Normal | 23
  High | 80
  Low and high | 0
  Missing | 0

17. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Bilirubin, Creatinine, and Direct Bilirubin Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Bilirubin, creatinine, and direct bilirubin were measured in micromoles per liter (µmol/L).
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Bilirubin, low | 31
  Bilirubin, normal | 68
  Bilirubin, high | 4
  Bilirubin, low and high | 0
  Bilirubin, missing | 0
  Creatinine, low | 54
  Creatinine, normal | 49
  Creatinine, high | 0
  Creatinine, low and high | 0
  Creatinine, missing | 0
  Direct bilirubin, low | 0
  Direct bilirubin, normal | 4
  Direct bilirubin, high | 0
  Direct bilirubin, low and high | 0
  Direct bilirubin, missing | 99

18. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Calcium, Chloride, Glucose, Phosphate, Potassium, Sodium, and Urea Nitrogen Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Calcium, chloride, glucose, phosphate, potassium, sodium, and urea nitrogen were measured in millimoles per liter (mmol/L).
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Calcium, low | 0
  Calcium, normal | 84
  Calcium, high | 19
  Calcium, low and high | 0
  Calcium, missing | 0
  Chloride, low | 52
  Chloride, normal | 51
  Chloride, high | 0
  Chloride, low and high | 0
  Chloride, missing | 0
  Glucose, low | 13
  Glucose, normal | 86
  Glucose, high | 4
  Glucose, low and high | 0
  Glucose, missing | 0
  Phosphate, low | 0
  Phosphate, normal | 82
  Phosphate, high | 21
  Phosphate, low and high | 0
  Phosphate, missing | 0
  Potassium, low | 0
  Potassium, normal | 80
  Potassium, high | 23
  Potassium, low and high | 0
  Potassium, missing | 0
  Sodium, low | 8
  Sodium, normal | 93
  Sodium, high | 1
  Sodium, low and high | 1
  Sodium, missing | 0
  Urea nitrogen, low | 2
  Urea nitrogen, normal | 86
  Urea nitrogen, high | 15
  Urea nitrogen, low and high | 0
  Urea nitrogen, missing | 0

19. Secondary Outcome: CT Period: Number of Participants With a Worst Abnormal Post-Baseline Creatinine Clearance Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. Creatinine clearance was measured in milliliters per minute per 1.73 square meters of body surface area (mL/min/1.73 m^2).
Time Frame: up to Week 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
Participants
  Low | 0
  Normal | 2
  High | 4
  Low and high | 0
  Missing | 97

20. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline ALT, ALP, AST, CL, and LDH Value of Low, Normal, High, Low and High, and Missing
Description: Low: participants with ≥1 low value but not any high values. High: participants with ≥1 high value but not any low values. Normal: participants without any low or high values. Low and high: participants with both low and high values. ALT, ALP, AST, CK, and LDH were measured in units per liter.
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  ALT, low | 5
  ALT, normal | 78
  ALT, high | 5
  ALT, low and high | 0
  ALT, missing | 4
  ALP, low | 14
  ALP, normal | 69
  ALP, high | 5
  ALP, low and high | 0
  ALP, missing | 4
  AST, low | 2
  AST, normal | 82
  AST, high | 4
  AST, low and high | 0
  AST, missing | 4
  CK, low | 5
  CK, normal | 56
  CK, high | 27
  CK, low and high | 0
  CK, missing | 4
  LDH, low | 9
  LDH, normal | 72
  LDH, high | 7
  LDH, low and high | 0
  LDH, missing | 4

21. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Albumin Value of Low, Normal, High, Low and High, and Missing
Description: as for outcome 16
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Low | 0
  Normal | 19
  High | 69
  Low and high | 0
  Missing | 4

22. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Bilirubin, Creatinine, and Direct Bilirubin Value of Low, Normal, High, Low and High, and Missing
Description: as for outcome 17
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Bilirubin, low | 40
  Bilirubin, normal | 43
  Bilirubin, high | 5
  Bilirubin, low and high | 0
  Bilirubin, missing | 4
  Creatinine, low | 58
  Creatinine, normal | 30
  Creatinine, high | 0
  Creatinine, low and high | 0
  Creatinine, missing | 4
  Direct bilirubin, low | 0
  Direct bilirubin, normal | 4
  Direct bilirubin, high | 0
  Direct bilirubin, low and high | 0
  Direct bilirubin, missing | 88

23. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Calcium, Chloride, Glucose, Phosphate, Potassium, Sodium, and Urea Nitrogen Value of Low, Normal, High, Low and High, and Missing
Description: as for outcome 18
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Calcium, low | 2
  Calcium, normal | 72
  Calcium, high | 14
  Calcium, low and high | 0
  Calcium, missing | 4
  Chloride, low | 54
  Chloride, normal | 34
  Chloride, high | 0
  Chloride, low and high | 0
  Chloride, missing | 4
  Glucose, low | 12
  Glucose, normal | 72
  Glucose, high | 4
  Glucose, low and high | 0
  Glucose, missing | 4
  Phosphate, low | 1
  Phosphate, normal | 62
  Phosphate, high | 25
  Phosphate, low and high | 0
  Phosphate, missing | 4
  Potassium, low | 1
  Potassium, normal | 66
  Potassium, high | 21
  Potassium, low and high | 0
  Potassium, missing | 4
  Sodium, low | 17
  Sodium, normal | 70
  Sodium, high | 0
  Sodium, low and high | 1
  Sodium, missing | 4
  Urea nitrogen, low | 4
  Urea nitrogen, normal | 65
  Urea nitrogen, high | 19
  Urea nitrogen, low and high | 0
  Urea nitrogen, missing | 4

24. Secondary Outcome: LTS Period: Number of Participants With a Worst Abnormal Post-Baseline Creatinine Clearance Value of Low, Normal, High, Low and High, and Missing
Description: as for outcome 19
Time Frame: from Week 9 up to Week 52 (44 weeks)
Population: LTS Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92
Participants
  Low | 0
  Normal | 10
  High | 11
  Low and high | 0
  Missing | 71

25. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Weeks 8, 44, and 52
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 8, 44, and 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
millimeters of mercury (mmHg)
  Baseline, SBP | 112.7 (11.14)
  Change from Baseline at Week 8, SBP: number analyzed (Participants) | 95
  Change from Baseline at Week 8, SBP | 0.6 (10.01)
  Change from Baseline at Week 44, SBP: number analyzed (Participants) | 69
  Change from Baseline at Week 44, SBP | -1.4 (11.10)
  Change from Baseline at Week 52, SBP: number analyzed (Participants) | 69
  Change from Baseline at Week 52, SBP | 1.0 (10.77)
  Baseline, DBP | 71.0 (8.03)
  Change from Baseline at Week 8, DBP: number analyzed (Participants) | 95
  Change from Baseline at Week 8, DBP | 0.2 (8.35)
  Change from Baseline at Week 44, DBP: number analyzed (Participants) | 69
  Change from Baseline at Week 44, DBP | 0.1 (9.31)
  Change from Baseline at Week 52, DBP: number analyzed (Participants) | 69
  Change from Baseline at Week 52, DBP | 1.0 (8.04)

26. Secondary Outcome: Change From Baseline in Pulse at Weeks 8, 44, and 52
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 8, 44, and 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
beats per minute
  Baseline | 78.8 (12.71)
  Change from Baseline at Week 8: number analyzed (Participants) | 95
  Change from Baseline at Week 8 | 0.5 (11.23)
  Change from Baseline at Week 44: number analyzed (Participants) | 69
  Change from Baseline at Week 44 | -0.6 (11.69)
  Change from Baseline at Week 52: number analyzed (Participants) | 69
  Change from Baseline at Week 52 | -0.4 (12.18)

27. Secondary Outcome: Change From Baseline in Respiration Rate at Weeks 8, 44, and 52
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 8, 44, and 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
breaths per minute
  Baseline | 16.1 (2.50)
  Change from Baseline at Week 8: number analyzed (Participants) | 95
  Change from Baseline at Week 8 | 0.7 (6.91)
  Change from Baseline at Week 44: number analyzed (Participants) | 69
  Change from Baseline at Week 44 | -0.5 (1.91)
  Change from Baseline at Week 52: number analyzed (Participants) | 69
  Change from Baseline at Week 52 | -0.1 (1.88)

28. Secondary Outcome: Change From Baseline in Body Temperature at Weeks 8, 44, and 52
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 8, 44, and 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
degrees Celsius
  Baseline | 36.5 (0.42)
  Change from Baseline at Week 8: number analyzed (Participants) | 95
  Change from Baseline at Week 8 | 0.0 (0.40)
  Change from Baseline at Week 44: number analyzed (Participants) | 69
  Change from Baseline at Week 44 | 0.1 (0.43)
  Change from Baseline at Week 52: number analyzed (Participants) | 69
  Change from Baseline at Week 52 | 0.1 (0.44)

29. Secondary Outcome: Change From Baseline in Height at Weeks 8 and 52
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 8 and 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
centimeters
  Baseline | 165.1 (9.88)
  Change from Baseline at Week 8: number analyzed (Participants) | 95
  Change from Baseline at Week 8 | 0.7 (1.20)
  Change from Baseline at Week 52: number analyzed (Participants) | 68
  Change from Baseline at Week 52 | 3.1 (3.31)

30. Secondary Outcome: Change From Baseline in Weight at Weeks 8 and 52
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 8 and 52
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103
kilograms
  Baseline | 65.0 (18.25)
  Change from Baseline at Week 8: number analyzed (Participants) | 95
  Change from Baseline at Week 8 | 0.9 (3.11)
  Change from Baseline at Week 52: number analyzed (Participants) | 68
  Change from Baseline at Week 52 | 3.8 (7.01)

31. Secondary Outcome: Plasma Concentration of Ruxolitinib
Description: Blood samples were drawn to assess plasma concentration.
Time Frame: prior to study cream application at Weeks 2 and 4
Population: Pharmacokinetic (PK) Population: all participants who applied ruxolitinib cream at least once and provided at least 1 postbaseline PK sample (1 PK measurement). Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nM)
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 100
nanomoles per liter (nM)
  Week 2: number analyzed (Participants) | 92
  Week 2 | 21.4 (27.7)
  Week 4: number analyzed (Participants) | 88
  Week 4 | 24.6 (38.2)

ADVERSE EVENTS:
Time Frame: from the time of Informed Consent Form signing until at least 30 days after the last application of study drug (up to approximately 20 months)
Description: Adverse events were assessed in members of the Full Analysis Set, comprised of all participants who applied ruxolitinib cream at least once.
Arm/Group | Ruxolitinib 1.5% Cream BID
All-Cause Mortality (participants affected / at risk) | 0/103
Serious Adverse Events (participants affected / at risk) | 2/103
Other Adverse Events (participants affected / at risk) | 20/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib 1.5% Cream BID (N=103)
Depression (Psychiatric disorders) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib 1.5% Cream BID (N=103)
Nasopharyngitis (Infections and infestations) | 9 (13)
Upper respiratory tract infection (Infections and infestations) | 11 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT05456529/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT05456529/SAP_001.pdf